CLINICAL TRIAL: NCT06656988
Title: A Contrast Medium Sparing Strategy Using Automated Carbon Dioxide Injection During PERIpheral Vascular Interventions for PREVENTion of Major Adverse Kidney Events (MAKE): the PeriPREVENT Randomized Controlled Trial
Brief Title: A Contrast Medium Sparing Strategy Using Automated CO2 Injection During PVI for Prevention of Major Adverse Kidney Events (MAKE)
Acronym: PeriPREVENT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Sabine Steiner, Prof. Dr., University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PeriPREVENT; 2024-512876-37-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-16; First posted 2024-10-24 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Peripheral Vascular Diseases; Kidney Diseases
Keywords: carbon dioxide; contrast medium; iodinated contrast medium; CA-AKI; angiography; angioplasty
MeSH Terms: conditions — Peripheral Vascular Diseases; Kidney Diseases | interventions — Carbon Dioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard angiography using iodinated Contrast Medium (CM) (Active Comparator): For patients randomised in the control group, a planned infrainguinal peripheral vascular intervention (PVI, not subject to the trial) will be performed with iso-osmolar or low-osmolar iodinated CM as contrast agent.
  The trial sites may use iodinated CM as defined per local routine. In line with current recommendations , the use of high-osmolar CM will be prohibited in the trial.
  Interventions: Drug: Iodinated Contrast Media (ICM)
- Contrast medium sparing strategy using CO2 injection as contrast agent, bailout option iodinated CM (Experimental): For patients randomised in the intervention group, a planned infrainguinal peripheral vascular intervention (PVI, not subject to the trial) will be performed with CO2 as contrast agent.
  For the CO2 injection the Angiodroid® Injector will be used according to the recent user manual. The use of the Angiodroid® system allows a fully automatic injection with digital control. Automatic CO2 injection enhances patient tolerability as the gas injection is performed in a less explosive, more controlled manner.
  Iodinated CM (as described in the above section) is used as bailout option in case of inadequate image quality or intraprocedural intolerance of CO2 angiography by the patient. The reasons for use and the amount of CM must be carefully recorded.
  Interventions: Drug: CO2

INTERVENTIONS:
Drug: CO2 — CO2 will be used as contrast medium sparing strategy during peripheral angiography
  Other Names: carbon dioxide
  Arms: Contrast medium sparing strategy using CO2 injection as contrast agent, bailout option iodinated CM
Drug: Iodinated Contrast Media (ICM) — Iodinated contrast medium will be used as in routine care during peripheral angiography
  Arms: Standard angiography using iodinated Contrast Medium (CM)

SUMMARY:
The primary objective of the trial is to evaluate if an iodinated contrast medium sparing strategy using automated Carbon Dioxide (CO2) Injection prevents Major Adverse Kidney Events up to 90 days (MAKE90) in patients at moderately elevated risk for contrast-associated acute kidney injury (CA-AKI) undergoing infrainguinal peripheral vascular interventions (PVI).

DETAILED DESCRIPTION:
PeriPREVENT is a prospective, multi-centre, controlled, open-label, 1:1 randomized superiority trial with two parallel groups.

In the intervention group patients will undergo a routine peripheral angiographic intervention (PVI) using a maximally contrast medium sparing strategy with an automated CO2 injection system including iodinated CM as bailout option in case of insufficient image quality or patient's intolerability of CO2 angiography.

The control intervention is routine PVI using iodinated contrast media (CM) as standard of care.

All patients are followed up until 12 months after the PVI.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic peripheral arterial disease presenting with either acute symptoms (Rutherford clinical categories I-IIb) and/or chronic symptoms (Rutherford clinical categories 3-6)
2. Planned peripheral vascular intervention of infrainguinal arteries due to femoropopliteal and/or infrapopliteal lesions
3. Increased risk of CA-AKI identified by a baseline risk score of ≥ 5 points based on a published dedicated PVI risk score and a pre-angiographic estimated glomerular filtration rate (eGFR) < 60 ml/min/1.73 m²
4. Both angiographic strategies seem feasible at the investigator's discretion
5. Age 18 years or older
6. Written informed consent

Exclusion Criteria:

1. Very agitated patients
2. Patients with planned full anaesthesia during procedure
3. Patients with a life-expectancy less than one year
4. Patients confined to bed that are completely non-ambulatory
5. Known acute renal failure or known unstable renal function as evidenced by a recent increase in serum creatinine (SCr) of > 0.5 mg/dl or > 25% within 7 days
6. Iodinated contrast medium exposure within 7 days prior to procedure with change in SCr ≥ 0.1 mg/dl on two SCr measures ≥ 24 h apart
7. Advanced chronic kidney disease (CKD) with an eGFR < 30 ml/min/1.73m² and/or dialysis
8. Current use of nephrotoxic agents (aminoglycoside antibiotics, sulfonamides, amphotericin B, or pentamidine), or an active chemotherapy agent
9. Acute or chronic pulmonary disease requiring oxygen therapy
10. Patients with known patent foramen ovale or atrial septal defect
11. Patients with planned nitrous oxide anaesthesia during intervention
12. Patients with manifest hyperthyroidism or manifest thyrotoxicosis
13. Known allergies or hypersensitivity to iodinated contrast media that cannot be adequately pre-treated prior to index procedure
14. Patients with decompensated heart failure
15. Patients with manifest tetany
16. Planned further procedure with a need for > 10 ml of iodinated contrast medium (CM) in any location (e.g., CT scan, coronary angiography) within a period of 90 days
17. Any surgical procedure (except minor amputations) or intervention performed within 30 days prior to or planned within 90 days post index procedure
18. Fertile women (within two years of their last menstruation) without appropriate contraceptive measures (implanon, injections, oral contraceptives, intrauterine devices, partner with vasectomy) until day 30 after PVI.
19. Participation in other interventional trials. Exceptions are described in the trial protocol.
20. Suspected lack of compliance
21. Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1960 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
MAKE 90 | From the day of the peripheral vascular intervention (day 0) to day 90
  major adverse kidney events

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Steiner, Prof Dr, Principal Investigator — University Leipzig
Locations (9):
- Austria (2):
  - Tirol Kliniken Innsbruck, Innsbruck
  - Universitätsklinik für Innere Medizin II, Vienna
- Germany (7):
  - Kreiskrankenhaus Alsfeld, Alsfeld
  - Universitäts-Herzzentrum Freiburg-Bad Krozingen, Bad Krozingen
  - MVZ CCB Frankfurt und Main-Taunus GbR, Frankfurt a.M.
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum rechts der Isar der Technischen Universität München, München
  - MEDINOS Kliniken des Landkreises Sonneberg GmbH, Sonneberg
  - GRN - Klinik Weinheim, Weinheim

IPD SHARING:
Plan to Share IPD: Yes
After publication of the major results and upon reasonable request from researchers performing an individual patient data meta-analysis, individual patient data that underlie published results will be shared after de-identification. This requires approval by the local Institutional Review Board (IRB) of the researcher requesting the data along with public registration of the meta-analysis.
  Summary statistics that go beyond the scope of published material will be made available to researchers for meta-analysis upon reasonable request and if the necessary data analysis is not unduly time-consuming. Together with publication of the main results, the statistical analysis plan will be made publicly available. The trial protocol will be published in a medical journal as soon as possible after approval of the trial.
Supporting Information: Study Protocol
Time Frame: The study protocol is made publicly available with the approval via CTIS.
Access Criteria: Please contact the coordinating investigator.